CLINICAL TRIAL: NCT04117945
Title: A Randomized Phase II Study of Regorafenib Followed by Anti-EGFR Monoclonal Antibody Therapy Versus the Reverse Sequencing for Metastatic Colorectal Cancer Patients Previously Treated With Fluoropyrimidine, Oxaliplatin and Irinotecan (REVERCE II)
Brief Title: Regorafenib, With Cetuximab or Panitumumab, for the Treatment of Unresectable, Locally Advanced, or Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-1809; NCI-2019-06518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-1809 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: BRAF V600E Negative; KRAS Gene Mutation Negative; Locally Advanced Unresectable Colorectal Adenocarcinoma; Metastatic Colorectal Adenocarcinoma; NRAS Gene Mutation Negative; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; Panitumumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (regorafenib) (Experimental): Patients receive regorafenib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If received as initial treatment, patients who experience disease progression may switch over to the other treatment regimen, per treating physician discretion.
  Interventions: Drug: Regorafenib
- Arm B (cetuximab, panitumumab, irinotecan) (Experimental): Patients receive cetuximab or panitumumab IV over 30-90 minutes on days 1 and 15. Patients may also receive irinotecan IV on days 1 and 15 as determined by the study doctor. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If received as initial treatment, patients who experience disease progression may switch over to the other treatment regimen, per treating physician discretion.
  Interventions: Biological: Cetuximab; Drug: Irinotecan; Biological: Panitumumab

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm B (cetuximab, panitumumab, irinotecan)
Drug: Irinotecan — Given IV
  Arms: Arm B (cetuximab, panitumumab, irinotecan)
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
  Arms: Arm B (cetuximab, panitumumab, irinotecan)
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Stivarga
  Arms: Arm A (regorafenib)

SUMMARY:
This phase II trial how well regorafenib and anti-EGFR therapy (cetuximab or panitumumab) works for the treatment of patients with colorectal cancer that cannot be removed by surgery (unresectable), has spread to nearby tissue or lymph nodes (locally advanced), or has spread to other places in the body (metastatic). Regorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab or panitumumab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. The purpose of this research study is to compare the effects, good and/or bad, of taking regorafenib follow by cetuximab or panitumumab, to those that receive cetuximab or panitumumab before regorafenib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the overall survival between evaluable patients who were randomized to receive regorafenib followed by anti-EGFR monoclonal antibody therapy compared to those that receive anti-EGFR monoclonal antibody followed by regorafenib.

SECONDARY OBJECTIVES:

I. To compare the first progression free survival (PFS1) of patients between evaluable patients who were randomized to receive regorafenib followed by anti-EGFR monoclonal antibody therapy compared to those that receive anti-EGFR monoclonal antibody followed by regorafenib II. To compare the second progression free survival (PFS2) of patients between evaluable patients who were randomized to receive regorafenib followed by anti-EGFR monoclonal antibody therapy compared to those that receive anti-EGFR monoclonal antibody followed by regorafenib.

III. To compare the sequential treatment progression free survival (stPFS) of patients between evaluable patients who were randomized to receive regorafenib followed by anti-EGFR monoclonal antibody therapy compared to those that receive anti-EGFR monoclonal antibody followed by regorafenib.

IV. To assess the frequency and severity of adverse events between evaluable patients who were randomized to receive regorafenib followed by anti-EGFR monoclonal antibody therapy compared to those that receive anti-EGFR monoclonal antibody followed by regorafenib.

V. To compare the objective response rate (ORR), while on initial treatment, between evaluable patients who were randomized to receive regorafenib followed by anti-EGFR monoclonal antibody therapy compared to those that receive anti-EGFR monoclonal antibody followed by regorafenib VI. To compare the objective response rate (ORR), while on sequential treatment, between evaluable patients who were randomized to receive regorafenib followed by anti-EGFR monoclonal antibody therapy compared to those that receive anti-EGFR monoclonal antibody prior to regorafenib.

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess plasma pharmacodynamics biomarkers of response and resistance to therapy.

II. To explore any correlation between tissue and blood based biomarkers and clinical outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive regorafenib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Per the treating physician's discretion, patients who experience disease progression may initiate a treatment regimen consisting of cetuximab or panitumumab intravenously (IV) over 30-90 minutes on days 1 and 15. Patients may also receive irinotecan IV on days 1 and 15 as determined by the study doctor. Cycles repeat every 28 days until disease progression or unacceptable toxicity.

ARM B: Patients receive cetuximab or panitumumab IV over 30-90 minutes on days 1 and 15. Patients may also receive irinotecan IV on days 1 and 15 as determined by the study doctor. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Per the treating physician's discretion, patients who experience disease progression may initiate a treatment regimen consisting of regorafenib PO QD on days 1-21. Cycles repeat every 28 days until disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months for up to 3 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, unresectable distant metastatic or locally advanced colorectal adenocarcinoma
* KRAS, NRAS wild type
* BRAF v600E wildtype
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Life expectancy of >= 3 months per estimation of treating physician
* Absolute neutrophil count (ANC) >= 1200/mm^3 (obtained =< 7 days prior to randomization)
* Platelet count >= 75,000/mm^3 (obtained =< 7 days prior to randomization)
* Hemoglobin >= 9.0 g/dL (obtained =< 7 days prior to randomization)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 7 days prior to randomization)
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer) (obtained =< 7 days prior to randomization)
* Serum creatinine =< 1.5 x ULN (obtained =< 7 days prior to randomization)
* International normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.5 x ULN (obtained =< 7 days prior to randomization)

  * NOTE: Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care
* Alkaline phosphatase limit =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement of their cancer) (obtained =< 7 days prior to randomization)
* Negative serum pregnancy test done =< 7 days prior to randomization for women of childbearing potential only.

  * NOTE: Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test. The definition of adequate contraception will be based on the judgment of the treating physician
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Disease progression on or intolerable to any of the following: fluoropyrimidine, oxaliplatin and irinotecan
* Able to swallow and retain oral medication
* Willing to provide tissue and blood samples for correlative research purposes
* Willing to allow transfer of tissue and blood samples, clinical information, and outcome data collected from this trial for future research

Exclusion Criteria:

* Prior treatment with regorafenib, cetuximab or panitumumab
* Major surgical procedure, open biopsy, or significant traumatic injury =< 28 days prior to randomization
* Congestive heart failure > New York Heart Association (NYHA) class 2.

  * NOTE: Class 3 is defined as marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g., walking short distances (20-100m). They are comfortable at rest. Class 4 is defined as patients with severe limitations. Experiences symptoms even while at rest. Mostly bed bound
* Unstable angina (angina symptoms at rest), new-onset angina (begun =< 3 months prior to randomization) or myocardial infarction =< 6 months prior to randomization
* Cardiac arrhythmias requiring anti-arrhythmic therapy. Note: Pace makers, beta blockers or digoxin are permitted
* Uncontrolled hypertension. (Systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management)
* History of or current pheochromocytoma
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism =< 6 months prior to randomization
* Ongoing infection > grade 2 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0
* Known history of chronic hepatitis B or C
* Patients with seizure disorder requiring medication
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of randomization and is clinically stable with respect to the tumor at the time of randomization. Note: Patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies)
* History of organ allograft (including corneal transplant)
* Evidence or history of bleeding diathesis or any hemorrhage or bleeding event > CTCAE v5.0 grade 3 =< 4 weeks prior to randomization
* Non-healing wound, ulcer, or bone fracture
* Substance abuse, medical, psychological or social conditions that may interfere with the patient?s participation in the study or evaluation of the study results
* High-frequency microsatellite instability (MSI-H) patients who have not received prior PD-1 monoclonal antibody (mAb) therapy
* Concurrent anti-cancer therapy =< 3 weeks from randomization (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization)
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* History of known persistent proteinuria of CTCAE v5.0 grade 3 or higher (>= 3.5 g/24 hrs)
* Any malabsorption condition
* Unresolved toxicity greater than CTCAE v5.0 grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity =< grade 2
* Albumin levels < 2.5 g/dl
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
  * NOTE: Men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form (ICF) until at least 3 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the treating physician, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known history of human immunodeficiency virus (HIV) infection or active hepatitis B or C infection requiring treatment with antiviral therapy
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer =< 3 years prior to randomization EXCEPT for cervical cancer in-situ, treated ductal carcinoma in situ of the breast, curatively treated nonmelanoma skin carcinoma, noninvasive aerodigestive neoplasms, or superficial bladder tumor (Ta [Non-invasive tumor], Tis [carcinoma in situ] and T1 [Tumor invades lamina propria]). Note: All cancer treatments for cancers that were distinct in a primary site other than colorectal must be completed at least 3 years prior to randomization (i.e., signature date of the informed consent form)
* Pleural effusion or ascites that causes respiratory compromise (>= CTCAE v5.0 grade 2 dyspnea)
* Any condition which, in the treating physician?s opinion, makes the subject unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2025-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Ahn, Principal Investigator — Academic and Community Cancer Research United
Locations (15):
- United States (15):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Regorafenib): Patients receive regorafenib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If received as initial treatment, patients who experience disease progression may switch over to the other treatment regimen, per treating physician discretion.
  >
  > Regorafenib: Given PO
- Arm B (Cetuximab, Panitumumab, Irinotecan): Patients receive cetuximab or panitumumab IV over 30-90 minutes on days 1 and 15. Patients may also receive irinotecan IV on days 1 and 15 as determined by the study doctor. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If received as initial treatment, patients who experience disease progression may switch over to the other treatment regimen, per treating physician discretion.
  >
  > Cetuximab: Given IV
  >
  > Irinotecan: Given IV
  >
  > Panitumumab: Given IV
Period: Overall Study
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Started | 12 | 10
Crossed Over to Other Treatment | 4 | 8
Completed | 0 | 0
Not Completed | 12 | 10
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Disease Progression | 0 | 2
Not completed — Ineligible | 8 | 7

BASELINE CHARACTERISTICS:
Population: Only eligible patients were included in analysis
Groups:
- Arm A (Regorafenib): Patients receive regorafenib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If received as initial treatment, patients who experience disease progression may switch over to the other treatment regimen, per treating physician discretion.>
  > Regorafenib: Given PO
- Arm B (Cetuximab, Panitumumab, Irinotecan): Patients receive cetuximab or panitumumab IV over 30-90 minutes on days 1 and 15. Patients may also receive irinotecan IV on days 1 and 15 as determined by the study doctor. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If received as initial treatment, patients who experience disease progression may switch over to the other treatment regimen, per treating physician discretion.>
  > Cetuximab: Given IV>
  > Irinotecan: Given IV>
  > Panitumumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (8.19) | 54.0 (19.16) | 63.4 (15.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.6 (0.92) | 27.0 (3.52) | 24.5 (3.20)
Primary Tumor Site [Count of Participants; unit: Participants]
  Right | 4 | 3 | 7
  Left | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction>
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work>
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours>
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours>
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair>
  5. Dead
  Participants
    0 | 2 | 2 | 4
    1 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The median OS and 95% confidence intervals in each arm will be reported.
Time Frame: 20 months
Population: Only eligible patients were included in analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Number analyzed (Participants) | 4 | 3
months | 3.6 [0.7 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events. | 13.3 [7.9 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events.
Statistical Analysis 1: Comparison: Arm A (Regorafenib) vs Arm B (Cetuximab, Panitumumab, Irinotecan); Test type: Superiority; p = 0.8874, One-sided unstratified log-rank

2. Secondary Outcome: First Progression-free Survival (PFS)
Description: The median first PFS and 95% confidence intervals in each arm will be reported.
Time Frame: 11 months
Population: Only eligible patients were included in analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Number analyzed (Participants) | 4 | 3
months | 1.2 [0.7 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events. | 7.0 [3.9 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events.
Statistical Analysis 1: Comparison: Arm A (Regorafenib) vs Arm B (Cetuximab, Panitumumab, Irinotecan); Test type: Superiority; p = 0.9683, One-sided unstratified log-rank

3. Secondary Outcome: Second PFS
Description: The median second PFS and 95% confidence intervals in each arm will be reported.
Time Frame: 3 months
Population: Only patients that were eligible and experienced at least one progression were included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Number analyzed (Participants) | 2 | 2
months | 2.3 [NA to NA] — The limits of the confidence interval were not able to be estimated due to a low number of events. | 1.8 [1.8 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events.
Statistical Analysis 1: Comparison: Arm A (Regorafenib) vs Arm B (Cetuximab, Panitumumab, Irinotecan); Test type: Superiority; p = 0.0448, One-sided unstratified log-rank

4. Secondary Outcome: Sequential Treatment PFS
Description: The median PFS while on sequential treatment and 95% confidence intervals in each arm will be reported.
Time Frame: 12 months
Population: Only eligible patients were included in analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Number analyzed (Participants) | 4 | 3
months | 3.6 [0.7 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events. | 8.9 [5.9 to NA] — The upper limit of the confidence interval was not able to be estimated due to a low number of events.
Statistical Analysis 1: Comparison: Arm A (Regorafenib) vs Arm B (Cetuximab, Panitumumab, Irinotecan); Test type: Superiority; p = 0.9007, One-sided unstratified log-rank

5. Secondary Outcome: Objective Response Rate
Description: Point estimates and the corresponding 95% confidence intervals for the true success proportions in each arm will be reported.
Time Frame: 20 months
Population: Only eligible patients were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

6. Secondary Outcome: Sequential Treatment Objective Response Rate
Description: Point estimates and the corresponding 95% confidence intervals for the true success proportions will be reported.
Time Frame: 20 months
Population: Only patients that started sequential treatment were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

7. Secondary Outcome: Number of Patients Experiencing Adverse Events
Description: The number of patients who experience a grade 3 or higher adverse event (Common Terminology Criteria for Adverse Events [CTCAE] version [v.] 5.0), regardless of attribution, will be reported by arm.
Time Frame: 20 months
Population: Only eligible patients were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan)
Number analyzed (Participants) | 4 | 3
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 20 months
Groups:
- Crossover From Arm A: Regorafenib followed by anti-EGFR mAb
- Crossover From Arm B: Anti-EGFR mAb followed by regorafenib
Arm/Group | Arm A (Regorafenib) | Arm B (Cetuximab, Panitumumab, Irinotecan) | Crossover From Arm A | Crossover From Arm B
All-Cause Mortality (participants affected / at risk) | 4/12 | 6/10 | 2/4 | 6/8
Serious Adverse Events (participants affected / at risk) | 6/12 | 4/10 | 1/4 | 1/8
Other Adverse Events (participants affected / at risk) | 12/12 | 9/10 | 4/4 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Regorafenib) (N=12) | Arm B (Cetuximab, Panitumumab, Irinotecan) (N=10) | Crossover From Arm A (N=4) | Crossover From Arm B (N=8)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Regorafenib) (N=12) | Arm B (Cetuximab, Panitumumab, Irinotecan) (N=10) | Crossover From Arm A (N=4) | Crossover From Arm B (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 5 (13) | 3 (5) | 3 (3)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 8 (35) | 2 (4) | 5 (11)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 2 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (8) | 5 (16) | 1 (1) | 3 (6)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (9) | 1 (1) | 2 (2)
Fatigue (General disorders) | 10 (16) | 8 (40) | 3 (6) | 5 (13)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial throm time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (11) | 7 (13) | 2 (3) | 3 (4)
Alkaline phosphatase increased (Investigations) | 3 (4) | 6 (16) | 1 (9) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 7 (13) | 6 (17) | 2 (3) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (4) | 2 (3) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 3 (9) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (3) | 1 (3) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 2 (4) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 4 (7) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 6 (23) | 1 (8) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (9) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6) | 2 (2) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 7 (16) | 4 (12) | 2 (17) | 5 (12)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 2 (10) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6) | 6 (29) | 2 (19) | 4 (8)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (11) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (17) | 6 (21) | 2 (8) | 5 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT04117945/Prot_SAP_000.pdf